CLINICAL TRIAL: NCT01496924
Title: Swallowing Rehabilitation of Dysphagic Tracheostomized Patients Under Mechanical Ventilation at Intensive Care Unit
Brief Title: Swallowing Rehabilitation of Dysphagic Tracheostomized Patients Under Mechanical Ventilation at ICU
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Katia Alonso Rodrigues, principal investigator, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP1802/06
Record Dates: First submitted 2011-11-21; First posted 2011-12-21 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Dysphagia
Keywords: Dysphagia; Intensive care units; Deglutition disorders; Rehabilitation
MeSH Terms: conditions — Deglutition Disorders | interventions — Speech Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- speech therapy group (Other): All dysphagic patients will be submitted to speech therapy
  Interventions: Other: speech therapy

INTERVENTIONS:
Other: speech therapy — A single oral-motor technique will be used in a 10-times series intercalated with rest. Swallowing training techniques comprised indirect therapy (swallowing of saliva) and direct therapy (swallowing of food).

SUMMARY:
There is an association between increased risk of oropharyngeal dysphagia and artificial ventilation through endotracheal tube, followed by tracheostomy. The aim of the present study is to analyze the outcomes of an early swallowing rehabilitation program of dysphagic tracheostomized patients under mechanical ventilation at the intensive care unit.

DETAILED DESCRIPTION:
This prospective study will be conduct in seven intensive care units of the university public hospital Inclusion criteria are: patients under mechanical ventilation and tracheostomy for at least 48 hours, appropriate level of consciousness (Glasgow coma scale ≥ 11), hemodynamic stability without need for vasoactive drugs; minimum mechanical ventilation parameters characterized by: pressure support ventilation (PSV) ≤ 20 cm H2O, positive end-expiratory pressure (PEEP) ≤ 8 cm H2O, fraction of inspired oxygen (FiO2) ≤ 50 and respiratory rate ≤ 30 inspirations per minute. Primary exclusion criteria are: patients who underwent surgery with resection of structures of oral cavity, pharynx, larynx and/or esophagus; nasal fracture or skull base fracture preventing otorhinolaryngological exam; possible surgical treatment after ICU admission with no reasonable time for carrying out the planned intervention; degenerative diseases characterized by outbreaks and remissions; past history of oropharyngeal dysphagia, previous speech therapy, excessive amount of thick tracheal secretion requiring frequent tracheal suctioning, end-stage of chronic obstructive pulmonary disease, tracheoesophageal fistula, allergy to dyes, and low survival expectancy.

The study consist of three stages: (1) sample selection with a test of the speaking valve and initial assessments, (2) swallowing rehabilitation and (3) post-treatment reassessments. Clinical assessments will be performed by speech-pathologists and otorhinolaryngologists with patients under mechanical ventilation. Subsequently, patients with dysphagia will be submitted to a rehabilitation program with standardized intervention, followed by a new assessment of abnormalities. The efficacy of swallowing treatment will be assessed by comparing the scores before and after treatment. Paired Student's test or Wilcoxon-test will be applied, according to data distribution. Categorical variables will be expressed as number and percentage and analyzed through McNemar test. All p-values will be two-sided and a p-value < 0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* admission in an ICU
* mechanical ventilation and tracheostomy for at least 48 hours
* appropriate level of consciousness (Glasgow coma scale ≥ 11)
* hemodynamic stability without need for vasoactive drugs
* minimum mechanical ventilation parameters characterized by pressure support ventilation (PSV) ≤ 20 cm H2O, positive end-expiratory pressure (PEEP) ≤ 8 cm H2O, fraction of inspired oxygen (FiO2) ≤ 50 and respiratory rate ≤ 30 inspirations per minute.

Exclusion Criteria:

* surgery with resection of structures of oral cavity, pharynx, larynx and/or esophagus
* nasal fracture or skull base fracture preventing otorhinolaryngological exam
* possible surgical treatment after ICU admission with no reasonable time for carrying out the planned intervention
* degenerative diseases characterized by outbreaks and remissions
* past history of oropharyngeal dysphagia
* previous speech therapy
* excessive amount of thick tracheal secretion requiring frequent tracheal suctioning
* end-stage of chronic obstructive pulmonary disease
* tracheoesophageal fistula
* allergy to dyes
* low survival expectancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
dysphagia improvement | participants will be followed for the duration of ICU stay, an expected average of 2 weeks"
  Otorhinolaryngological assessment will be carried out before and after treatment by means of a bedside video nasal endoscopic examination of swallowing, and included the evaluation of the following aspects: mobility of vocal folds, saliva and food swallowing, swallowing trigger time, food stasis in pharyngeal recesses, laryngeal penetration, tracheal aspiration, pharyngeal clearance after swallowing, laryngeal sensitivity and cough reflex, both by the speech-language pathologist and the otorrhinolaryngologist

CONTACTS AND LOCATIONS:
Overall Officials: Katia Alonso, PHD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Intensive Care Unit - Hospital Sao Paulo, São Paulo, São Paulo, Brazil